CLINICAL TRIAL: NCT02650102
Title: The Role of miR-30 Family Dysregulation in Response to Antipsychotic Treatment
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Yong Xu, Dr Yong Xu, Shanxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 81571319
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Olanzapine; Quetiapine Fumarate; Aripiprazole; ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- antipsychotics (Experimental): This group was treated with one of 5 antipsychotics(risperidone/olanzapine/aripiprazole/quetiapine/ziprasidone) randomly.
  Interventions: Drug: Risperidone; Drug: Olanzapine; Drug: Quetiapine; Drug: Aripiprazole; Drug: Ziprasidone
- health control (No Intervention): This group was treated with no invention

INTERVENTIONS:
Drug: Risperidone — a kind of antipsychotics
  Other Names: Risperdal
  Arms: antipsychotics
Drug: Olanzapine — a kind of antipsychotics
  Other Names: Zyprexa
  Arms: antipsychotics
Drug: Quetiapine — a kind of antipsychotics
  Other Names: Seroquel
  Arms: antipsychotics
Drug: Aripiprazole — a kind of antipsychotics
  Other Names: Abilifya
  Arms: antipsychotics
Drug: Ziprasidone — a kind of antipsychotics
  Other Names: Geodon
  Arms: antipsychotics

SUMMARY:
The aberrant expression of micro-RNAs (miRNAs) has been described in many human diseases, including schizophrenia (SZ). The previous work has indicated a strong genetic association between the miRNA-30e precursor (pre-miR-30e) and the risk of SZ. However, to date, few reports have focused on the expression level of the miR-30 family (miR-30s) and its networks of co-regulation in SZ, even in response to antipsychotic treatment. Given this, the investigator first constructed a hybrid miRNA-TF (transcription factor)-gene-PPI (protein-protein interactions) network focusing on miR-30s by bioinformatics technology. The investigator then selected several candidate miR-30s and key regulators for further validation. These candidates were then quantified by real-time quantitative PCR (qRT-PCR) in an independent cohort of 200 healthy controls and 200 drug-free SZ patients, among which were followed up by 12-week antipsychotic treatment. Furthermore, the investigator evaluated the correlation between the change in gene expression and the improvement of symptoms.

DETAILED DESCRIPTION:
Schizophrenia is one of the most serious mental disorder，which is characterized by high prevalence rate ,high recurrence rate, could increase patients' disability and burden of disease. But the pathological mechanism is so far unknown. Until recently, more attention are focused on gene dysregulation hypothesis. The preliminary works of our laboratory prompted that microRNA-30e gene polymorphism and expression abnormal may be related to schizophrenia. Combined with previous studies showed that miRNA disorder involved in neurodevelopmental obstacle and neuropsychiatric disease, the investigators surmised: miR-30e dysregulation can impact the occurrence and development of schizophrenia. This study will carry on the multidimensional research by using the technology of neurobiology, molecular genetics,neuroimaging and so on, and integrate methods of molecular, cell, animal and human body tracking, so as to:(1) Explaining the transcription and regulation mechanisms of target genes of miR-30e,and building the gene regulatory network of schizophrenia as the core of miR-30e.(2)To investigate the pathogenesis of miR-30e participate in schizophrenia, and to evaluate the clinical value of miR-30e in peripheral blood on the disease diagnose, genotyping, predicting efficacy and ending. The object of this study is to provide new scientific data and research ideas for further exploring the neurobiological basis of schizophrenia, and recognize pathophysiological mechanisms of schizophrenia, ultimately to improve and strengthen the new situation in schizophrenia prevention.

ELIGIBILITY:
Inclusion Criteria:

* Unrelated Han Chinese recruited from the north of China.
* Drug-free for at least one month before enrollment.
* Clinical diagnosis of schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) criteria for SZ (American Psychiatric Association, 1994), relying on the Chinese Version of the Modiﬁed Structured Clinical Interview for DSM-IV TR Axis I Disorders Patient Edition (SCID-I/P,11/2002 revision).

Exclusion Criteria:

* Pregnant or had signiﬁcant medical conditions.
* Unstable psychiatric features (e.g., suicidal feelings).
* A history of substance abuse or drug addiction within the previous 6 months, with the exception of nicotine dependence.
* Other Axis I co-morbid disorders were not excluded.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of schizophrenics with antipsychptic treatment who achieved remission assessed by PANSS. | Number of schizophrenics with 12-week antipsychptic treatment who achieved remission assessed by PANSS.
  The clinical effects were assessed by trained and experienced psychiatrists with the Positive and Negative Syndrome Scale (PANSS) before and after 12-week treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Xu, Doctor, Principal Investigator — Shanxi Medical University
Locations (1):
- First Clinical Medical College of Shanxi Medical University, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: Yes